CLINICAL TRIAL: NCT02041767
Title: Assessment of Prostatic Tissue Concentration of Ertapenem After a Pre-operative Administration
Acronym: ERTAPRO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P090205
Record Dates: First submitted 2014-01-20; First posted 2014-01-22 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Benign Prostatic Hyperplasia (BPH) Requiring Surgical Resection
Keywords: Ertapenem; prostatic diffusion; antibioprophylaxy; pharmacokinetics; benign prostatic hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Ertapenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- group A (Experimental): One single perfusion of 1g of ertapenem 1 hour prior to prostate surgical resection
  Interventions: Drug: Ertapenem
- group B (Experimental): One single perfusion of 1g of ertapenem 12 hour prior to prostate surgical resection
  Interventions: Drug: Ertapenem

INTERVENTIONS:
Drug: Ertapenem — One single injection of 1g of ertapenem before surgery

SUMMARY:
The purpose of this study is to demonstrate the prostatic diffusion in significant concentration of ertapenem achieved after a pre-operative single administration.

DETAILED DESCRIPTION:
Ertapenem is an antibiotic belonging to carbapenems family and used in infections with Gram-negative bacilli with extended spectrum beta lactamase (ESBL). Its efficacy has been demonstrated in abdominal, soft tissue, pulmonary, skin and gynaecological infections. Recently it has been compared to ceftriaxone in urinary infections demonstrating his efficacy and tolerance.

The purpose of this study is to assess its benefit in probabilistic strategy by demonstrating its prostatic diffusion in significant concentration when administrated in a pre-operative single injection.

Patients were divided in two groups receiving a single injection of 1g of ertapenem 1h or 12h before endoscopic surgery of prostate hyperplasia.

Concentration of ertapenem was measuring on blood sample and on chips resection of prostate during endoscopic surgery.

To demonstrate the prostatic diffusion in significant amount of ertapenem, the prostatic concentration of ertapenem had to be higher than the minimal inhibitory concentration (MIC) for 40% of the time of injection interval.

ELIGIBILITY:
Inclusion Criteria:

* Acceptance and understanding of the consent form (signed)
* 18-80 years old patients
* BPH needing endoscopic resection according to French Urology Association recommendations
* Procedure and follow up made in investigator center
* normal digital rectal examination
* PSA :
* patient > 69 years old, not necessary
* patient < 69 years old, PSA<20 and if 4<PSA<20, the ratio free PSA/total PSA must be >10%
* patient with renal clearance >60 estimated with MDRD
* patient affiliated to the social security

Exclusion Criteria:

* personal or familial history of prostatic or genito-urinary cancer
* personal history of pelvic irradiation
* personal history of hormone-therapy
* personal history of prostatic adenomectomy by abdominal approach
* personal history of allergy to beta-lactamines
* urinary tract infection or bacterial colonisation at the time of procedure
* carbapenems treatment in the two weeks before surgery
* hyperresponsivness to ertapenem or other carbapenems antibiotic
* patient with renal clearance estimated with MDRD <60
* patient with catheter or probe permanently

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-01 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Prostatic concentration of ertapenem | at the time of surgery
  To observe whether a significant intra-prostatic concentration of ertapenem can be obtained after a pre-operative single administration.

SECONDARY OUTCOMES:
Prostatic concentration of ertapenem | at the time of surgery
  To observe the difusion of ertapenem by comparing 1h versus12h injection prior to surgery

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Lortholary, Md, PhD, Study Chair — Service de Maladies Infectieuses et Tropicales, Hôpital Necker, 149 rue de Sèvres; Marc-Olivier Timsit, Md, PhD, Principal Investigator — Service d'Urologie, HEGP, 20 rue Leblanc, 75015 Paris, France.
Locations (1):
- HEGP Hospital, Paris, France

REFERENCES:
- [Background] Dariane C, Amin A, Lortholary O, Lalli A, Michel C, Le Guilchet T, Treluyer J, Nguyen-Khoa T, De Toma C, Urien S, Mejean A, Bourget P, Timsit M. Concentrations plasmatiques et intra-prostatiques d'ertapeneme apres administration preoperatoire : experience prospective monocentrique - etude ERTAPRO. Prog Urol. 2015 Nov;25(13):775. doi: 10.1016/j.purol.2015.08.121. No abstract available. French. PMID 26544316
- [Background] Dariane C, Amin A, Lortholary O, Lalli A, Michel C, Le Guilchet T, Treluyer JM, Nguyen-Khoa T, De Toma C, Urien S, Mejean A, Bourget P, Timsit MO. Plasma and intraprostatic concentrations of ertapenem following preoperative single dose administration: a single-centre prospective experience and clinical implications-the ERTAPRO study. Int J Antimicrob Agents. 2016 Aug;48(2):168-74. doi: 10.1016/j.ijantimicag.2016.04.027. Epub 2016 Jun 2. PMID 27324263
- [Background] Alhambra A, Cuadros JA, Cacho J, Gomez-Garces JL, Alos JI. In vitro susceptibility of recent antibiotic-resistant urinary pathogens to ertapenem and 12 other antibiotics. J Antimicrob Chemother. 2004 Jun;53(6):1090-4. doi: 10.1093/jac/dkh218. Epub 2004 Apr 29. PMID 15117925
- [Background] Tomera KM, Burdmann EA, Reyna OG, Jiang Q, Wimmer WM, Woods GL, Gesser RM; Protocol 014 Study Group. Ertapenem versus ceftriaxone followed by appropriate oral therapy for treatment of complicated urinary tract infections in adults: results of a prospective, randomized, double-blind multicenter study. Antimicrob Agents Chemother. 2002 Sep;46(9):2895-900. doi: 10.1128/AAC.46.9.2895-2900.2002. PMID 12183244
- [Background] Jimenez-Cruz F, Jasovich A, Cajigas J, Jiang Q, Imbeault D, Woods GL, Gesser RM; Protocol 021 Study Group. A prospective, multicenter, randomized, double-blind study comparing ertapenem and ceftriaxone followed by appropriate oral therapy for complicated urinary tract infections in adults. Urology. 2002 Jul;60(1):16-22. doi: 10.1016/s0090-4295(02)01664-3. PMID 12100914
- [Background] Wells WG, Woods GL, Jiang Q, Gesser RM. Treatment of complicated urinary tract infection in adults: combined analysis of two randomized, double-blind, multicentre trials comparing ertapenem and ceftriaxone followed by appropriate oral therapy. J Antimicrob Chemother. 2004 Jun;53 Suppl 2:ii67-74. doi: 10.1093/jac/dkh208. PMID 15150185